CLINICAL TRIAL: NCT06041932
Title: Pentoxifylline Plus Carvedilol vs Carvedilol Monotherapy in Preventing New Decompensation in Stable Cirrhotic Patients With Prior Decompensation, an Open Label Randomised Control Trial
Brief Title: Pentoxifylline Plus Carvedilol vs Carvedilol Monotherapy in Preventing New Decompensation in Stable Cirrhotic Patients With Prior Decompensation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-62
Record Dates: First submitted 2023-08-23; First posted 2023-09-18 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-08

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Carvedilol; Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentoxiphylline plus Carvedilol (Experimental): Pentoxiphylline plus Carvedilol
  Interventions: Drug: Carvedilol; Drug: Pentoxifylline
- Carvedilol (Active Comparator): PCarvedilol
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Drug: Carvedilol — Carvedilol
Drug: Pentoxifylline — Pentoxiphylline
  Arms: Pentoxiphylline plus Carvedilol

SUMMARY:
Cirrhotics with decompensation have increased risk of morbidity and mortality. There is increased portal pressure leading to decompensation. Carvedilol is a standard therapy given to cirrhotic patient with clinically significant portal hypertension to reduce portal pressure. Pentoxifylline is a nonspecific phosphodiesterase inhibitor with anti-inflammatory properties. It reduces portal hypertension, decreases lipopolysaccharide-induced liver injury, improves nonalcoholic steatohepatitis, prevents development of HRS in ascites and SAH, prevents hepatopulmonary syndrome. Investigator want to study whether addition of pentoxifylline to carvediolol vs carvedilol monotherapy reduces the risk of mortality and further decompensation in cirrhotics with prior decompensation.

DETAILED DESCRIPTION:
* Study population: Cirrhotic patients with prior decompensation at least 3 months ago
* Study design: A Open label randomized controlled trial
* Sample size Assuming decompensation in Arm 1 as 25%, and 10% in Arm 2, alpha error- 5, power - 80, 160 patients, 10 % lost to follow up - 180, Each arm 90 patients.
* Intervention Arm 1 : Carvedilol Arm 2 : Pentoxiphylline plus Carvedilol
* Monitoring and assessment

At enrollment:

* - Complete history and physical examination
* Prior ascites, Hepatic encephalopathy, acute variceal bleed.
* Time to prior decompensation
* Pattern and number of prior decompensation
* Prior spontaneous bacterial peritonitis, hydrothorax, Acute on chronic liver failure, acute kidney injury
* Use of Non selective beta blockers, norfloxaxin, rifaximin and albumin
* Recent herbal/drugs intake
* History of EVL or other endotherapy
* History of hypertension, diabetes mellitus
* Fever , signs of sepsis
* Examination- Sarcopenia, fraility, icterus, pedal edema

At follow-up (at 3 month, 6 month, 9 month, 12 month): Physical (preferably)

• Complete history and physical examination

* New onset ascites, Hepatic encephalopathy, acute variceal bleed, clinical Jaundice
* Time to new decompensation from enrollment
* Pattern and number of new decompensation
* Other complications - Spontaneous bacterial peritonitis, hydrothorax, Acute on chronic liver failure, acute kidney injury.
* Recent herbal/drugs intake
* History of EVL or other endotherapy
* Hypertension, Diabetes control
* Fever , signs of sepsis
* Examination- Sarcopenia, fraility, icterus, pedal edema, ascites, Hepatic encephalopathy

Clinical evaluation

* Etiology of chronic liver disease (Baseline)
* Control of etiological factor (Baseline, 3 monthly) Alcohol - No relapse, if relapse - severity HBV - on antivirals, HBV DNA -ve HCV - HCV RNA -ve Metabolic risk factors control- DM, HT, weight etc.
* Severity of liver disease (Baseline, 3 monthly) MELD score, MELD-Na score, CTP score
* Complications (at 3 month, 6 month, 9 month, 12 month):

Overt Hepatic Encephalopathy, Portal hypertension related bleed, clinical jaundice, ascites, hyponatremia, Acute kidney injury, spontaneous bacterial peritonitis, Infections

Laboratory parametres

* Baseline (at enrollment) - Blood : KFT, LFT, CBC, INR, AFP, TNF-a, IL-6, CRP, VWF, ADAM TS 13 Imaging : USG abdomen, LSM, SSM, ECHO Hemodynamics : HVPG (not mandatory)
* At 3 and 6 month - Blood : KFT, LFT, CBC, INR Imaging : USG abdomen, LSM, SSM
* At 1 year (end of follow-up) Blood : KFT, LFT, CBC, INR, AFP, TNF-a, IL-6, CRP, VWF, ADAM TS 13 Imaging : USG abdomen, LSM, SSM Hemodynamics : HVPG ( not mandatory)

  - STATISTICAL ANALYSIS:
* Data will be reported as mean + SD.
* Categorical variables will be compared using the chi-square test or Fisher exact test
* Normal continuous variables will be compared using the Student's t test
* Non normal continuous variables will be compared using the Mann-Whitney rank-sum test (unpaired data) or the Wilcoxon test (paired data).
* The actuarial probability of survival will be calculated by the Kaplan-Meier method and compared using the log-rank test.
* A Cox regression analysis will be performed to identify independent prognostic factors for survival.
* Univariate and multivariate analysis will be used whenever applicable. - Adverse effects Carvedilol - Bradycardia, hypotension, giddiness, diarrhea, insomnia, hyperglycemia, weight gain, increased BUN, increased nonprotein nitrogen (NPN), increased cough, abnormal vision.

Pentoxiphylline - Abdominal discomfort, bloating, diarrhea, Dizziness, headache, flushing, chest pain, arrhythmias, hypertension, dyspnea, tachycardia, and hypotension.

- Stopping rule If primary end point achieved or any adverse event due to drug

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years
2. Cirrhosis with prior clinical decompensation (ascites, Hepatic encephalopathy, Portal Hypertension related bleed)
3. No current clinical decompensation (for at least 3 months)

Exclusion Criteria:

1. Post TIPS/ BRTO/ SAE patients
2. Post renal or liver transplantation
3. History of CAD, ischemic cardiomyopathy, PVD, ventricular arrythmia
4. Presence of clinical ascites, HE, Jaundice
5. Last clinical decompensation within 3 months.
6. Ongoing significant alcohol use
7. Active HCV/HBV infection (Detectable HCV RNA/ HBV DNA)
8. Prior Intolerance to carvedilol and hypersensitivity to Pentoxyfylline
9. Use of Pentoxifylline within last 1 month
10. AIH/PBC
11. Lack of informed consent
12. Hepatocellular carcinoma / Portal vein thrombosis/ Budd Chiari Syndrome
13. Non-cirrhotic portal hypertension
14. Ongoing CAM/Hepatotoxic drug intake
15. Known HIV infection
16. Pregnant women
17. HepatoPulmonary Syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of New onset clinical decompensation (any of overt HE, variceal bleed, clinical jaundice and ascites) at 1 year in two groups. | 1 year

SECONDARY OUTCOMES:
Precipitants, timing of new-onset decompensation at 6 months in two groups. | 6 months
Mortality at 6 months | 6 months
Precipitants, timing of new-onset decompensation at 12 months in two groups | 12 months
Mortality at 12 months in two groups. | 12 months
Changes in Liver stiffness measured by Fibroscan at 6 months | 6 months
Changes in Liver stiffness measured by Fibroscan at 12 months | 12 months
Change in ESR at 6 months in both groups | 6 months
Change in CRP at 6 months in both groups | 6 months
Change in IL 6 at 6 months in both groups | 6 months
Change in TNF Alpha at 6 months in both groups | 6 months
Change in Von Willebrand factor at 6 months in both groups | 6 months
Change in ADAM TS 13 at 6 months in both groups | 6 months
Change in ESR at 12 months in both groups. | 12 months
Change in CRP at 12 months in both groups | 12 months
Change in IL 6 at 12 months in both groups | 12 months
Change in TNF Alpha at 12 months in both groups | 12 months
Change in Von Willebrand factor at 12 months in both groups | 12 months
Change in ADAM TS 13 at 12 months in both groups | 12 months
Dose of Pentoxifylline and Carvedilol at 6 months. | 6 months
Dose of Pentoxifylline and Carvedilol at 12 months | 12 months
Number of patients with change in CTP in both groups. | 3 month, 6 month, 9 month and at end of 1 year
Number of patients with change in MELD score in both groups. | 3 month, 6 month, 9 month and at end of 1 year
  MELD minimum value=6 and maximum value=40
Incidence of Hepatocellular carcinoma at 6 months between two groups. | 6 months
Incidence of Hepatocellular carcinoma at 12 months between two groups. | 12 months
Incidence of Portal vein thrombosis at 6 months between two groups. | 6 months
Incidence of Portal vein thrombosis at 12 months between two groups. | 12 months
Number of patients with adverse events in both the groups. | 6 months and 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences., New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No